CLINICAL TRIAL: NCT00517283
Title: A Study by Scintigraphy to Evaluate the Effect of Exenatide on Gastric Emptying in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H8O-EW-GWAM
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; gastric emptying; exenatide; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Exenatide 5 mcg - Exentatide 10 mcg - Placebo
  Interventions: Drug: exenatide and placebo
- Sequence 2 (Experimental): Exenatide 10 mcg - Placebo - Exenatide 5 mcg
  Interventions: Drug: Exenatide and placebo
- Sequence 3 (Experimental): Placebo - Exenatide 5 mcg - Exenatide 10 mcg
  Interventions: Drug: Exenatide and placebo

INTERVENTIONS:
Drug: exenatide and placebo — Period 1 = Subcutaneous injections of exenatide 5mcg twice daily for 4 days and once in the morning of the 5th day. Period 2 = Subcutaneous injections of exenatide 5mcg twice daily for 2 days, followed by 2 days of twice daily 10 mcg doses, 10mcg once in the morning of the 5th day. Period 3 = Subcutaneous injections of placebo in an amount equivalent to exenatide twice daily for 4 days and once in the morning of the 5th day. A washout of at least 2.5 days will occur between each treatment period.
  Other Names: Byetta; AC2993; synthetic exendin-4
  Arms: Sequence 1
Drug: Exenatide and placebo — Period 1 = Subcutaneous injections of exenatide 5mcg twice daily for 2 days, followed by 2 days of twice daily 10 mcg doses, 10mcg once in the morning of the 5th day. Period 2 = Subcutaneous injections of placebo in an amount equivalent to exenatide twice daily for 4 days and once in the morning of the 5th day. Period 3 = Subcutaneous injections of exenatide 5mcg twice daily for 4 days and once in the morning of the 5th day. A washout of at least 2.5 days will occur between each treatment period.
  Other Names: Byetta; AC2993; synthetic exendin-4
  Arms: Sequence 2
Drug: Exenatide and placebo — Period 1 = Subcutaneous injections of placebo in an amount equivalent to exenatide twice daily for 4 days and once in the morning of the 5th day. Period 2 = Subcutaneous injections of exenatide 5mcg twice daily for 4 days and once in the morning of the 5th day. Period 3 = Subcutaneous injections of exenatide 5mcg twice daily for 2 days, followed by 2 days of twice daily 10 mcg doses, 10mcg once in the morning of the 5th day. A washout of at least 2.5 days will occur between each treatment period.
  Other Names: Byetta; AC2993; synthetic exendin-4
  Arms: Sequence 3

SUMMARY:
As exenatide slows the rate at which materials leave the stomach, it is likely to alter the rate of intestinal absorption of oral drugs when administered within a certain timeframe relative to exenatide. In addition, the residence time within the stomach of other medication may be prolonged and data from this study will help assess the change in residence time in the presence of therapeutic doses of exenatide. This study will also evaluate the relationship between blood levels of exenatide and parameters measuring rate of stomach emptying.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least 1 year history of type 2 diabetes mellitus.
* Subjects controlled by oral antidiabetic agents or diet and exercise demonstrated by a screening HbA1c ≥7.0% and ≤10.0%.
* Between the body mass index (BMI) of 19 kg/m2 and 40 kg/m2, inclusive.

Exclusion Criteria:

* Within 4 months of the initial dose of study drug, have received a drug that has not received regulatory approval for any indication.
* Persons who have previously completed or withdrawn from this study or any other study investigating exenatide.
* Subjects who are using drugs that significantly affect gastrointestinal motility (including acarbose, metoclopramide, and macrolide antibiotics).
* Subjects who intend to start new concomitant medication during the study, including over-the counter medication, apart from occasional intake of paracetamol or vitamin/mineral supplements. Anti-emetic medication may be permitted at the investigator's discretion, except those that affect gastrointestinal motility.
* Subjects who have used insulin for more than 4 weeks within 3 months prior to screening.
* Blood donation of more than 500 mL in the last 3 months of screening or any blood donation within the last month.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To detect the mean difference in half gastric emptying time for a solid meal between any treatment and placebo | up to 12 hours post meal consumption
  A dose of exenatide or placebo is given before the morning meal. After eating the test meal, images will be recorded at approximately 5 minute intervals from ingestion of the test meal until 3 hours after the meal, then every 10 minutes until 6 hours after the meal. In cases where significant radioactivity is observed at 6 hours after the meal, additional scintigraphic images may be taken periodically at the discretion of the investigator, until counts approach low values for up to 12 hours after the meal.

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (1):
- Research Site, Nottingham, United Kingdom